CLINICAL TRIAL: NCT06438237
Title: Validation of a Prediction Model for Inadequate Bowel Preparation Before Colonoscopy Based on a Systematic Review and Meta-analysis
Brief Title: Validation of a Prediction Model for Inadequate Bowel Preparation
Status: Completed | Type: Observational
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Xingshun Qi, Director of Gastroenterology, General Hospital of Shenyang Military Region
Other Study IDs: V-PMIBP
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2024-05

CONDITIONS: Bowel Preparation; Colonoscopy
Keywords: Bowel preparation for colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Patients undergoing colonoscopy in General Hospital of Northern Theater Command: Patients were informed to eat semi-liquid and non-slag diet for breakfast and lunch and full-liquid diet for dinner on the day before colonoscopy, and be fasting on the day of colonoscopy. A split-dose 3 L PEG regimen was used for all patients.
  Interventions: Procedure: Bowel preparation before colonoscopy
- Patients undergoing colonoscopy in First Affiliated Hospital of China Medical University: Patients were informed to eat semi-liquid and non-slag diet for breakfast and lunch and full-liquid diet for dinner on the day before colonoscopy, and be fasting on the day of colonoscopy. A split-dose 2 L PEG regimen was used for all patients.
  Interventions: Procedure: Bowel preparation before colonoscopy
- Inpatients undergoing colonoscopy in Second Affiliated Hospital of Army Medical University: We retrospectively collect data of inpatients undergoing colonoscopy. Patients were informed to eat semi-liquid and non-slag diet for breakfast and lunch and full-liquid diet for dinner on the day before colonoscopy, and be fasting on the day of colonoscopy. A full-dose 3 L PEG regimen was used for all patients.
  Interventions: Procedure: Bowel preparation before colonoscopy
- Patients undergoing colonoscopy in No. 960 Hospital: Patients were informed to eat semi-liquid and non-slag diet for breakfast and lunch and full-liquid diet for dinner on the day before colonoscopy, and be fasting on the day of colonoscopy. Split-dose 3 L PEG, sodium phosphate or sodium picosulfate regimen were used according to the doctor's advice.
  Interventions: Procedure: Bowel preparation before colonoscopy

INTERVENTIONS:
Procedure: Bowel preparation before colonoscopy — Patients use purgative for bowel cleansing before colonoscopy.

SUMMARY:
We have developed a novel inadequate bowel preparation prediction model based on a systematic review and meta-analysis. The goal of this multicenter observational study is to validate the accuracy of this model.

DETAILED DESCRIPTION:
The primary outcome is quality of bowel preparation. The secondary outcomes include polyp/adenoma detection rate, willingness of undergoing colonoscopy again and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients (age is ≥18 years old);
2. patients undergoing colonoscopy;
3. written informed consent.

Exclusion Criteria:

1. patients undergoing emergent colonoscopy;
2. patients with major psychiatric disorders;
3. pregnant or breast feeding patients;
4. patients with contraindications for colonoscopy (e.g., heart failure, renal insufficiency);
5. patients suspected to have intestinal obstruction, stenosis or perforation;
6. poor compliance with the bowel preparation protocol (poor compliance is indicated if the dose of medication was < 75% of the prescribed dose;
7. incomplete colonoscopy because of other circumstances apart from inadequate cleansing
8. patients previously enrolled in this study.

Ages: 18 Years to 94 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing colonoscopy
Sampling Method: Probability Sample
Enrollment: 2360 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Quality of bowel preparation | During the procedure of colonoscopy
  A total BBPS score ≥6 with BBPS score ≥2 for each colon segment was considered to have adequate bowel preparation. Each segment of the colon is scored from 0 to 3, with higher scores indicating superior cleansing, and summed for a total score that can range from 0 to 9.

SECONDARY OUTCOMES:
Adenoma and/or polyp detection rate | During the procedure of colonoscopy
  Proportion of patients with at least one adenoma and/or polyp detected during colonoscopy
Number of polyps and/or adenomas | During the procedure of colonoscopy
  Number of polyps and/or adenomas detected during colonoscopy
Adverse events | Before the procedure of colonoscopy
  Incidence of abdominal pain, bloating, nausea/vomiting after intake of purgative.

CONTACTS AND LOCATIONS:
Overall Officials: Xingshun Qi, Principal Investigator — Department of Gastroenterology, General Hospital of Northern Theater Command
Locations (1):
- Department of Gastroenterology, General Hospital of Northern Theater Command (formerly called General Hospital of Shenyang Military Area), Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):620-5. doi: 10.1016/j.gie.2008.05.057. Epub 2009 Jan 10. PMID 19136102